CLINICAL TRIAL: NCT06236204
Title: Arthroscopic Scapholunate Ligament Reconstruction, Volar and Dorsal Reconstruction, as Treatment for Dysfunction of the Scapholunate Joint With Insufficiency of the Scapholunate Ligament and Secondary Stabilizers
Brief Title: Arthroscopic Scapholunate Ligament Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Regionaal Ziekenhuis Heilig Hart Tienen (Other)
Responsible Party: Principal Investigator, Goorens Chul Ki, orthopaedic surgeon, principal investigator, Regionaal Ziekenhuis Heilig Hart Tienen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RZ Tienen EC 109
Record Dates: First submitted 2023-01-25; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Scapholunate Dissociation
Keywords: scapholunate instability; reconstruction

STUDY DESIGN:
Intervention Model Description: prospective single center - single surgeon
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arthroscopic Scapholunate Ligament Reconstruction (Experimental): Experimental: patients with dynamic scapholunate instability wrist arthroscopy: bone-tendon reconstruction of the volar and dorsal part of the scapholunate complex
  Interventions: Procedure: Arthroscopic Scapholunate Ligament Reconstruction

INTERVENTIONS:
Procedure: Arthroscopic Scapholunate Ligament Reconstruction — reconstruction of the SL ligament with palmaris tendon graft tunneled through the scaphoid and lunate as described by Corella et al.

SUMMARY:
Arthroscopical reconstruction of the volar and dorsal part of the scapholunate ligament as treatment for complete scapholunate ligament injury, but reducible carpal malalignment.

This prospective study aims to evaluate the clinical and functional outcome of this technique on the short and middle term

DETAILED DESCRIPTION:
Classical arthroscopic techniques for scapholunate instability consist of debridement, thermal shrinkage, and percutaneous pinning. Good results are obtained in acute lesions or in chronic partial tears, but they are less predictable when the lesion is complete, because of the poor healing capacity of the scapholunate ligament and because it is not possible to perform an anatomic ligamentous reconstruction with these techniques. Open techniques are thus required for reconstruction, but they damage the soft tissues. Corella et al. published a description and cadaver study of an arthroscopic ligamentoplasty, trying to combine the advantages of arthroscopic techniques (minimally invasive surgery) and open techniques (reconstruction of the ligament). With this approach, it is possible to reconstruct the dorsal scapholunate ligament and the secondary stabilizers while causing minimal damage to the soft tissues and avoiding injury to the posterior interosseous nerve and detachment of the dorsal intercarpal ligament. Arthroscopic scapholunate volar and dorsal ligament reconstruction achieves an anatomic reconstruction to provide a strong construct for early mobilization.

ELIGIBILITY:
Inclusion Criteria:

* Scapholunate dysfunction, complete irrepairable lesion of the SL ligament and the secondary stabilizers (RSC-LRL-SRL) EWAS stage 4-5, no arthritis, with reducible malalignment
* 18 - 65 years

Exclusion Criteria:

* - associated lesions, fractures
* neurological disorder affecting the upper limb, history of wrist lesion involving the same wrist, dementia, substance abuse, severe psychiatric disorder and previous injured contralateral wrist

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
passive and active range of motion (degrees) operated and contralateral side | preop
  flexion, extension, ulnar and radial deviation
passive and active range of motion (degrees) operated and contralateral side | postoperative 3 months
  flexion, extension, ulnar and radial deviation
passive and active range of motion (degrees) operated and contralateral side | postoperative 6 months
  flexion, extension, ulnar and radial deviation
passive and active range of motion (degrees) operated and contralateral side | postoperative 12 months
  flexion, extension, ulnar and radial deviation
grip strength (kg) operated and contralateral side | preop
  dynamometer (kg)
grip strength (kg) operated and contralateral side | postoperative 3 months
  dynamometer (kg)
grip strength (kg) operated and contralateral side | postoperative 6 months
  dynamometer (kg)
grip strength (kg) operated and contralateral side | postoperative 12 months
  dynamometer (kg)
pain (visual analogue scale) | preop
  Visual analogue Scale (0 no pain -10 cm worst pain)
pain (visual analogue scale) | postoperative 3 months
  Visual analogue Scale Scale (0 no pain -10 cm worst pain)
pain (visual analogue scale) | postoperative 6 months
  Visual analogue Scale Scale (0 no pain -10 cm worst pain)
pain (visual analogue scale) | postoperative 12 months
  Visual analogue Scale (0 no pain -10 cm worst pain)
Disabilities of the Arm, Shoulder and Hand score | preop
  function score (0 is best -100 is worst)
Disabilities of the Arm, Shoulder and Hand score | postoperative 3 months
  function score (0 is best -100 is worst)
Disabilities of the Arm, Shoulder and Hand score | postoperative 6 months
  function score (0 is best -100 is worst)
Disabilities of the Arm, Shoulder and Hand score | postoperative 12 months
  function score (0 is best -100 is worst)

SECONDARY OUTCOMES:
patient satisfaction after treatment | postoperative 12 months
  visual analogue scale (0 is worst -10 cm is best)
complications | postoperative 12 months
  descriptive
arthroscopical assessment of the scapholunate stability | intraoperative
  according to European Wrist Arthroscopy Society classification (EWAS1 best -5 worst)
scapholunate distance, carpal angles | preop
  radiological follow-up (distance in mm or angles in degrees)
scapholunate distance, carpal angles | postoperative 12 months
  radiological follow-up (distance in mm or angles in degrees)

CONTACTS AND LOCATIONS:
Overall Officials: Kjell Van Royen, MD, Study Chair — Universitair Ziekenhuis Brussel
Locations (1):
- Department of orthopaedics RZ Tienen, Tienen, Belgium